CLINICAL TRIAL: NCT03048812
Title: Clinical Outcomes Using Different Attachment Types for Single-implant Mandibular Overdentures: a Crossover Clinical Trial
Brief Title: Attachment Types for Single-implant Mandibular Overdentures: a Crossover Clinical Trial
Acronym: SIMODA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Associate Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UFG_43585
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Edentulous Mouth; Complete Edentulism
Keywords: Dental implant; Mandibular overdenture; Cross-over study
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the AB sequence receive treatment A in the first period and treatment B in the second period, whereas experimental units that are randomized to the BA sequence receive treatment B in the first period and treatment A in the second period
Who Masked: Outcomes Assessor
Masking Description: The outcome assessment will be blinded for assessment which treatment (O-Ring \Equator) is provided
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O'Ring attachment (A) (Experimental): One arm of our research will receive O'Ring attachment for 3 months and after this period they will recieve the second attachment Equator for more 3 months
  Interventions: Device: O'Ring Attachment (A); Device: Equator Attachment (B)
- Equator attachment (B) (Experimental): The second arm of our research will receive Equator attachment for 3 months and after this period they will recieve the second attachement O Ring for more 3 months
  Interventions: Device: O'Ring Attachment (A); Device: Equator Attachment (B)

INTERVENTIONS:
Device: O'Ring Attachment (A) — Attachment A will be inserted in three months of follow up,followed by treatment B in a random order
  Other Names: O'ring (Neodent, Curitiba, Paraná, Brazil)
Device: Equator Attachment (B) — Attachment B will be inserted in three months of follow up,followed by treatment A in a random order
  Other Names: Equator (Neodent, Curitiba, Paraná, Brazil)

SUMMARY:
Dental implants are often the preferred treatment option and in some clinical scenarios they are considered the standard of care to restore missing or damaged teeth, due to the limitations of conventional treatments. For fully edentulous subjects, conventional tissue-supported dentures in some cases are associated with severe subjective complaints and difficult adaptation, mainly the mandibular denture, resulting in limited function and detrimental effects on oral health-related quality of life, especially for older patients. The use of implants to retain a mandibular denture (overdenture) has been recommended as a suitable and low-cost alternative to improve denture stability, with positive effects on oral comfort and function. The two-implant mandibular overdenture has been considered an effective design to achieve clinical benefits for patients. However, the main problem facing two-implant overdenture is the high cost of implantation and the relative complexity of the surgical intervention, so the use of a single midline implant to retain a mandibular overdenture was suggested as a more viable solution for reducing costs and complexity of treatment with similar benefits compared to solutions with higher number of implants. Nevertheless, there are few studies that compared the performance of different retention systems and their effects on patient-centered outcomes, such as satisfaction with the dentures, oral health-related quality of life, individual preferences and other subjective ratings of clinical outcomes. Thus, the aim of this randomized clinical trial with a crossover design is to investigate the changes in clinical and patient-reported outcomes following the use of different retention systems for a single implant-retained mandibular overdenture Hypothesis: it was hypothesized that clinical and patient-reported outcomes of a single-implant mandibular overdenture is dependent on the type of retention system, and patients have distinct preferences in relation to different attachments

DETAILED DESCRIPTION:
The absence of all natural teeth has negative effects on edentulous subjects' quality of life. It affects badly the masticatory muscles, chewing efficiency and digestive process, ability to speak clearly, psycho-social impacts related to esthetics and non-self-confidence and it is often associated with increasing risk for chronic systemic diseases.

In Brazil, tooth loss is still a public health problem with high prevalence and negative impacts on the lives of individuals, despite the possibility of control by means of preventive and rehabilitation technologies aimed at promoting oral health. The prevalence of tooth loss is 76.6% in the general population, with a median of 6 teeth lost for the population aged 15 or more years old. There is a high prevalence of edentulism in the 65-74 years age group for the maxilla (63.1%) and mandible (37.5%). Epidemiological data showed that there was an improvement in the oral health status of adults as the demand for dentures. However, the major problem is still concentrated in the population aged 65 to 74, who had an average caries index rate of 27.1 in 2010 (in 2003 the average was 27.8) with a predominance of component lost by decay. From 2003 to 2010, the proportion of elderly people who need dentures dropped from 24% to 23% and from 16% to 15% for those who need partial dentures.

Although treatments using implants are widely available, conventional complete dentures are still an important part of oral health care for edentulous individuals, mainly due to economic reasons. However, conventional complete dentures do not always achieve all treatment goals regarding patient satisfaction and function, as a number of edentulous patients have problems with their dentures related to retention and comfort during mastication and speech, especially for the mandibular denture.

The limitations of conventional dentures make the implant-supported mandibular overdenture be considered the preferred option for a number of edentulous elders. As stabilization by implants can increase denture retention and stability, improve masticatory efficiency and patient satisfaction. Furthermore, there are scientific evidences that it also contributes for prevention of bone resorption.

The mandibular overdenture retained by two implants has been recommended as the minimum standard of care for the edentulous mandible. However, these consensus reports consider that anything less is negligent care disregard who cannot afford two implants, so the main problem related to implant overdenture is higher financial costs compared to the conventional complete denture. This is inconsistent with treatment concepts for the elderly, which include simplicity and cost effectiveness as major requirements in treatment planning.

In recent years, the single-implant mandibular overdenture has been proposed as an alternative to more complex overdenture designs for the treatment of mandibular edentulism. This treatment approach is assumed to be simpler and less costly than both the fixed implant treatment and the overdenture retained by two implants. It is also considered a more feasible option for geriatric patient groups because of their diminished functional demands and the favorable local bone condition in the symphyseal region that ensures satisfactory primary implant stability.

A series of clinical studies showed satisfactory results of the single-implant mandibular overdenture treatment regarding patient satisfaction and quality of life measures, as well as other clinical and radiographic outcomes such as implant survival rate, marginal bone loss and longitudinal implant stability. Although these studies differed on the experimental design, use of different implant and retention systems, loading protocols and evaluation of distinct clinical outcomes, they agree that the use of a single implant to retain an overdenture results in marked improvements compared to the conventional treatment Attachment systems used for implant-retained overdentures are small interlocking devices which links the implant with the dentures and this offer many balanced solutions between functions and oral comfort. The attachment systems allow an improvement in masticatory function, bite forces, food selection and quality of life. The retention design can be classified as mechanical, friction fit or magnetic. There are various attachments available for the clinicians in the market today such as bar connections, ball attachments, magnets, rigid or non-rigid telescopic copings and stud attachments.

Clinical studies also reported complications related to the clinical performance of attachment systems used for single-implant mandibular overdentures. Loss of retention and matrix replacement was one of the most common maintenance events in single mandibular overdenture patients, although some studies reported no need for replacement in the long-term follow-up. Studies showed great variation on the incidence of matrix replacement, although no comparison of different types of retention systems and no time-to-event analysis were reported. No difference between the incidence of repair and adjustments of mandibular overdentures supported by 1 or 2 implants was observed.

The impact of different attachment types on patient satisfaction and quality of life is recognized as a critical outcome requiring further investigation. For single-implant mandibular overdentures, studies reported in their majority the use of ball-o'ring, magnet and stud attachment systems. However, no evidences of the superiority of one system over another are available, considering both patient-reported outcomes such as individual preferences, easy to handle and oral comfort; and technical criteria such as level of retention, longevity, retrievability and the need of adjustments and replacement.

This study will focus in improving patient health care quality, satisfaction and treatment outcomes as it is considered the golden goal for studying clinical benefits from treatments by comparing between different types of attachments for single-implant mandibular overdenture treatment. This will be an experimental study using a randomized clinical trial with a crossover design to test if clinical and patient-reported outcomes are dependent on the type of retention system, and if patients have distinct preferences about the tested attachments.

ELIGIBILITY:
Inclusion Criteria:

* Be completely edentulous, male or female with no age restrictions;
* Need replacement or confection of new complete dentures defined according to normative criteria and/or own demand;
* Have no contraindications for implant placement surgery (mainly related to uncontrolled systemic diseases such as diabetes and hypertension);
* Have enough bone volume in the mandibular midline area for installation of an implant without the need for augmentation procedures;
* be able to understand and answer to the questionnaires used in the study;
* agree to participate in this study by providing a written informed consent.

Exclusion Criteria:

* present signs that they will be uncompliant in the follow-up appointments;
* present local conditions that could directly influence stability and/or retention of the dentures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Patient preference | 3 months
  Patient satisfaction with the attachment connected to the single implant overdenture

SECONDARY OUTCOMES:
Abutment loosening incidence | 3 months
  Incidence of abutment replacement due to loss of retention
Patient satisfaction | 3 months
  Patient satisfaction with the attachment connected to the single implant overdenture
Need for replacement | 3 months
  Incidence of attachment replacement due to loss of retention

CONTACTS AND LOCATIONS:
Overall Officials: Claudio R Leles, Doctorate, Principal Investigator — UFG

IPD SHARING:
Plan to Share IPD: No